CLINICAL TRIAL: NCT01658735
Title: Electrical Stimulation for Chronic Non-specific Low Back Pain in a Working-Age Population: A 12-Week Double Blinded Randomized Controlled Trial
Brief Title: Comparison of Electrotherapies for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Electronic Waveform Lab, Inc. (Industry)
Responsible Party: Principal Investigator, Matt Hughes, MD, MPH, Assistant Professor (clinical), University of Utah
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB_00052918; IRB_00052918
Record Dates: First submitted 2012-07-30; First posted 2012-08-07 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-02

CONDITIONS: Non-specific Chronic Low Back Pain
Keywords: Chronic low back pain; Electrotherapy; H-Wave; H wave; TENS; Trial
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- H-Wave Device (Active Comparator): H-Wave Device with Usual Care
  Interventions: Device: H-Wave
- TENS (Active Comparator): Transcutaneous electrical nerve stimulation (TENS) Device with Usual Care
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation (TENS)
- Sham Electrotherapy (Sham Comparator): Sham Device plus Usual Care.
  Interventions: Device: Sham

INTERVENTIONS:
Device: H-Wave — Proprietary electrotherapy device using electrical stimulation of unique wave form and energy level that is delivered through transcutaneous electrodes to nerves and soft tissue for analgesic effect.
  Other Names: H-Wave is the proprietary name of the device. There is only one model currently.
  Arms: H-Wave Device
Device: Transcutaneous Electrical Nerve Stimulation (TENS) — Electrotherapy device that delivers current at different frequency, amplitude, and wave form through cutaneous electrodes placed near body parts with pain for temporary analgesic effect. The study device is installed inside the same housing as the H-Wave Device and Sham Device, so that all appear the same. There are no identifying marks on the case that participants will recognize in order to maintain blinding.
  Other Names: Chattanooga Intellect TENS Device
  Arms: TENS
Device: Sham — The sham device is a TENS unit modified to have minimal electrical output. The device is installed in the same housing as the two active arms with equal weight, so that each device in the study appears identical.
  Arms: Sham Electrotherapy

SUMMARY:
The intent of this project is to execute a high-quality double-blinded randomized controlled clinical trial that compares the H-Wave® device with a commonly used TENS device with a sub-therapeutic electrocurrent device. This study will provide a definable level of evidence for treatment efficacy, and provide a basis for evidence-based recommendation for or against utilization for these two modalities. The results for H-Wave® device, if positive, could significantly impact morbidity by providing a non-invasive, non-pharmacologic treatment for symptomatic relief, and reduce overall disability and health care costs associated with chronic low back pain.

DETAILED DESCRIPTION:
H-Wave® Device Stimulation (Intervention A) plus usual care, transcutaneous electrical nerve stimulation (TENS) (Intervention B) plus usual care, and sham electrotherapy plus usual care (control). Each treatment arm will have identical participants enrolled (n=38 per arm) of with the same number of visits and investigator contact time.

Eligible participants will be allocated through computerized randomization utilizing a stratified permuted-block randomization employing random block sizes. Allocation is concealed. Participants and assessors will be blinded. Participants will not be told what types of electrotherapy devices are being studied, only that there are different types, and that they may be randomized to receive a sham device.

Patients will be instructed on the use of the device they received to perform daily home therapy. Subjects will be assessed at week 1, 4, 8 and 12 for the primary and secondary outcomes measures. Compliance to treatment will be measured through an electronic meter on each of the devices, as well as by patient diary. Patients will be allowed to receive usual care from their own health care provider, with the exception of invasive procedures or surgery. Results will be analyzed by intention to treat methods.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Low Back Pain of at least 3 months duration
* ages 18-65
* Current VAS Pain Rating of 5 on 10 point scale
* No pain below the knee
* 75% of pain located in low back or buttock pain rather than lower extremity pain
* Proficient in English
* Able to complete and tolerate treatment for the study period.

Exclusion Criteria:

* Prior home use of H-Wave Device or TENS.
* Prior history of spinal fusion or failed spinal surgery syndrome.
* Laminectomy, laminotomy or discectomy within 12 months of enrollment.
* Diagnostic or interventional injections or any low back surgeries not mentioned above, including radiofrequency, neuroablation within 6 months of enrollment.
* Current implanted cardiac demand pacemakers, defibrillators, cardiac pumps, or other implanted electronic devices.
* Active psychiatric disorders will be excluded (e.g. use of antipsychotic medication, bipolar disorder, schizophrenia, uncontrolled depression or anxiety disorder).
* Patients currently or who become pregnant will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2012-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Hughes, Principal Investigator — DFPM-ADMINISTRATION

REFERENCES:
- [Background] Thiese MS, Hughes M, Biggs J. Electrical stimulation for chronic non-specific low back pain in a working-age population: a 12-week double blinded randomized controlled trial. BMC Musculoskelet Disord. 2013 Mar 28;14:117. doi: 10.1186/1471-2474-14-117. PMID 23537462

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | H-Wave Device | TENS | Sham Electrotherapy
Started | 39 | 36 | 38
Completed | 34 | 29 | 34
Not Completed | 5 | 7 | 4
Not completed — Lack of Efficacy | 1 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | H-Wave Device | TENS | Sham Electrotherapy | Total
Number analyzed (Participants) | 39 | 36 | 38 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (12.1) | 48.5 (11.5) | 45.5 (12.0) | 47.6 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 16 | 41
  Male | 23 | 27 | 22 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 3
  Not Hispanic or Latino | 38 | 36 | 36 | 110
  Unknown or Not Reported | 0 | 0 | 0 | 0
Number of participants currently working at enrollment [Number; unit: participants]
  Yes | 29 | 28 | 31 | 88
  No | 10 | 8 | 7 | 25
Number of participants who have ever seen a Chiropractor for LBP [Number; unit: participants]
  Yes | 23 | 23 | 25 | 71
  No | 16 | 13 | 13 | 42
Number of participants who have seen a Physician for their current LBP [Number; unit: participants]
  Yes | 23 | 28 | 27 | 78
  No | 16 | 8 | 11 | 35
Number of participants who have been to a chronic pain clinic for their current LBP [Number; unit: participants]
  Yes | 5 | 5 | 1 | 11
  No | 34 | 31 | 37 | 102
Participants of participants who have ever had a MRI for their current LBP [Number; unit: participants]
  Yes | 17 | 17 | 17 | 51
  No | 22 | 19 | 21 | 62
Number of participants that have ever smoked greater than 100 cigarettes - lifetime [Number; unit: participants]
  Yes | 9 | 4 | 9 | 22
  No | 30 | 32 | 29 | 91
Number of participants who have ever seen a physical therapist for LBP [Number; unit: participants]
  Yes | 17 | 18 | 22 | 57
  NO | 22 | 18 | 16 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Oswestry Disability Index at 1 Week
Description: Measure of the change in Oswestry Disability Index (ODI) after one week of treatment compared with baseline measure.
  The ODI is a commonly used outcome-measure questionnaire for low back pain. It is a self-administered questionnaire divided into ten sections designed to assess limitations of various activities of daily living. Each section is scored on a 0-5 scale, 5 representing the greatest disability. The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage, with a possible range of 0 to 100. Higher scores represent higher reported disability.
Time Frame: 1 week
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | H-Wave Device | TENS | Sham Electrotherapy
Number analyzed (Participants) | 39 | 36 | 38
units on a scale | -2.507 [-4.56 to -0.45] | -4.725 [-6.94 to -2.51] | -4.752 [-6.94 to -2.56]

2. Primary Outcome: Change From Baseline in Oswestry Disability Index at 4 Weeks
Description: Measure of the change in Oswestry Disability Index (ODI) after four weeks of treatment compared with baseline measure.
  The ODI is a commonly used outcome-measure questionnaire for low back pain. It is a self-administered questionnaire divided into ten sections designed to assess limitations of various activities of daily living. Each section is scored on a 0-5 scale, 5 representing the greatest disability. The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage, with a possible range of 0 to 100. Higher scores represent higher reported disability.
Time Frame: Week 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | H-Wave Device | TENS | Sham Electrotherapy
Number analyzed (Participants) | 39 | 36 | 38
units on a scale | -5.002 [-7.51 to -2.5] | -5.135 [-7.88 to -2.39] | -4.581 [-7.25 to -1.91]

3. Primary Outcome: Change From Baseline in Oswestry Disability Index at 8 Weeks
Description: Measure of the change in Oswestry Disability Index (ODI) after eight weeks of treatment compared with baseline measure.
  The ODI is a commonly used outcome-measure questionnaire for low back pain. It is a self-administered questionnaire divided into ten sections designed to assess limitations of various activities of daily living. Each section is scored on a 0-5 scale, 5 representing the greatest disability. The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage, with a possible range of 0 to 100. Higher scores represent higher reported disability.
Time Frame: Week 8
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | H-Wave Device | TENS | Sham Electrotherapy
Number analyzed (Participants) | 39 | 36 | 38
units on a scale | -5.299 [-8.19 to -2.41] | -5.135 [-7.88 to -2.39] | -4.679 [-7.41 to -1.89]

4. Primary Outcome: Change From Baseline in Oswestry Disability Index at 12 Weeks
Description: Measure of the change in Oswestry Disability Index (ODI) after twelve weeks of treatment compared with baseline measure.
  The ODI is a commonly used outcome-measure questionnaire for low back pain. It is a self-administered questionnaire divided into ten sections designed to assess limitations of various activities of daily living. Each section is scored on a 0-5 scale, 5 representing the greatest disability. The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage, with a possible range of 0 to 100. Higher scores represent higher reported disability.
Time Frame: Week 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | H-Wave Device | TENS | Sham Electrotherapy
Number analyzed (Participants) | 39 | 36 | 38
units on a scale | -5.388 [-8.47 to -2.3] | -6.907 [-10.32 to -3.49] | -5.612 [-8.82 to -2.4]

5. Secondary Outcome: Change From Baseline in VAS Pain Score at 1 Week
Description: Measure of the change in visual analogue scale (VAS) after one week of treatment compared with baseline VAS measure.
  The VAS is a commonly used continuous scale measure for low back pain. For pain intensity, the scale is anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 10). Higher scores represent higher reported pain.
Time Frame: Week 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | H-Wave Device | TENS | Sham Electrotherapy
Number analyzed (Participants) | 39 | 36 | 38
units on a scale | -1.458 [-2.21 to -0.93] | -1.929 [-2.75 to -1.11] | -2.042 [-2.84 to -1.25]

6. Secondary Outcome: Change From Baseline in VAS Pain Score at 4 Weeks
Description: Measure of the change in visual analogue scale (VAS) after four weeks of treatment compared with baseline VAS measure.
  The VAS is a commonly used continuous scale measure for low back pain. For pain intensity, the scale is anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 10). Higher scores represent higher reported pain.
Time Frame: Week 4
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | H-Wave Device | TENS | Sham Electrotherapy
Number analyzed (Participants) | 39 | 36 | 38
units on a scale | -2.017 [-2.9 to -1.13] | -1.691 [-2.66 to -0.72] | -1.843 [-2.79 to -0.9]

7. Secondary Outcome: Change From Baseline in VAS Pain Score at 8 Weeks
Description: Measure of the change in visual analogue scale (VAS) after eight weeks of treatment compared with baseline VAS measure.
  The VAS is a commonly used continuous scale measure for low back pain. For pain intensity, the scale is anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 10). Higher scores represent higher reported pain.
Time Frame: Week 8
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | H-Wave Device | TENS | Sham Electrotherapy
Number analyzed (Participants) | 39 | 36 | 38
units on a scale | -2.510 [-3.53 to -1.49] | -2.147 [-3.28 to -1.02] | -2.467 [-3.41 to -1.52]

8. Secondary Outcome: Change From Baseline in VAS Pain Score at 12 Weeks
Description: Measure of the change in visual analogue scale (VAS) after twelve weeks of treatment compared with baseline VAS measure.
  The VAS is a commonly used continuous scale measure for low back pain. For pain intensity, the scale is anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 10). Higher scores represent higher reported pain.
Time Frame: Week 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | H-Wave Device | TENS | Sham Electrotherapy
Number analyzed (Participants) | 39 | 36 | 38
units on a scale | -2.624 [-3.53 to -1.72] | -1.922 [-2.91 to -0.93] | -2.467 [-3.41 to -1.52]

ADVERSE EVENTS:
Time Frame: Within 12 weeks the participant was enrolled
Arm/Group | H-Wave Device | TENS | Sham Electrotherapy
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/36 | 0/38
Other Adverse Events (participants affected / at risk) | 2/39 | 2/36 | 1/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | H-Wave Device (N=39) | TENS (N=36) | Sham Electrotherapy (N=38)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Increase in Lower Extremity Tingling/Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Exacerbation of Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain/Flank pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Participant enrollment was based on chronic pain VAS score of >= 5.0 (0-10 scale). High baseline VAS scores did not translate to a priori hypothesized high ODI scores, resulting in study being underpowered to detect differences in primary outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No